CLINICAL TRIAL: NCT02944630
Title: Psychotherapy for Patients With Psoriasis: Effects in Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-PSO-2016-72
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Psoriasis
Keywords: quality of life; psychotherapy; psoriasis; treatments
MeSH Terms: conditions — Psoriasis | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: (Experimental): Receiving psychotherapy and medical treatment.
  Interventions: Behavioral: Psychotherapy
- Control (No Intervention): Awaiting group: Receiving medical treatment.

INTERVENTIONS:
Behavioral: Psychotherapy — Individual psychotherapy
  Arms: Experimental:

SUMMARY:
The aim of this study is to determine the benefits of individual psychotherapy on quality of life for people with psoriasis receiving medical treatment versus a control group (awaiting group) treated with medical treatment, without psychotherapy.

DETAILED DESCRIPTION:
Further investigations studies are needed to determine the efficacy of psychological interventions for people with psoriasis. The aim of this study is to determine the benefits of individual psychotherapy on quality of life for people with psoriasis receiving medical treatment versus a control group (awaiting group) treated with medical treatment, without psychotherapy.

This is an experimental randomized trial with control group. Quality of life, symptoms:

pruritus, scaling and pain, distress and the illness will be measured before and after the intervention using psychological and quality of life questionnaires, and dermatological evaluations for 120 subjects.

The investigators expect that the experimental group scores at the end of the psychotherapy program will be less than 4 points in Visual Analog Scale (VAS) for pruritus, scaling and pain. The Dermatology Quality of Life Index (DQLI) expected to be less than 4 points from the initial score, and the patients are expected to present less than 7 points in Hospital Anxiety and Depression Scale (HADS). The experimental group scores will be less than the control group for quality of life, symptoms and distress.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years old at the time of selection.
* Subjects diagnosed with moderated or severe psoriasis.
* Subjects with a ≥ 10 punctuation in DLQI questionnaire.
* Subjects that are in dermatological treatment.
* Patients should be able to understand and communicate with the investigator.

Exclusion Criteria:

* Subjects suffering from a serious concomitant illness.
* Subjects with a mental illness.
* Subjects who are performing psychiatric treatment.
* Subjects who are performing psychotherapy sessions both individual and group.
* Patients who have alcohol dependence or drug abuse.
* Subjects that present legal incapacity or limited legal capacity.
* Subjects presenting illiteracy or language barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Dermatology Quality of Life Index (DLQI) | 1 year
  The Dermatology Life Quality Index or DLQI, developed in 1994, was the first dermatology-specific Quality of Life instrument. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions in over 80 countries and is available in over 90 languages. Its use has been described in over 1000 publications including many multinational studies. The DLQI is the most frequently used instrument in studies of randomised controlled trials in dermatology.

SECONDARY OUTCOMES:
Visual analog scale (VAS) for pruritus | 1 year
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Operationally a VAS is usually a horizontal line, 100 mm in length. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Visual analog scale (VAS) for pain | 1 year
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Operationally a VAS is usually a horizontal line, 100 mm in length. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Visual analog scale (VAS) for scaling | 1 year
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Operationally a VAS is usually a horizontal line, 100 mm in length. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Hospital Anxiety and Depression Scale (HADS) | 1 year
  Hospital Anxiety and Depression Scale (HADS) was originally developed by Zigmond and Snaith (1983) and is commonly used by doctors to determine the levels of anxiety and depression that a patient is experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.
Psoriasis Area Severity Index (PASI) | 1 year
  The Psoriasis Area Severity Index (PASI) is an index used to express the severity of psoriasis. It combines the severity (erythema, induration and desquamation) and percentage of affected area.
Static Physician's Global Assessment (sPGA) | 1 year
  The PGA is a 5 point ordinal rating ranging from "clear" to "very severe psoriasis".
Body surface area (BSA) | 1 year
  The Body surface area is defined as 9% coverage for the head and neck, each arm, anterior and posterior leg as well as the four trunk quadrants respectively, leaving 1% for the genitalia. The BSA can also be estimated by the number of patients' hand areas affected, assuming that one "handprint" reflects approximately 1% of BSA

CONTACTS AND LOCATIONS:
Overall Officials: Esther Margarit de Miguel, Msc, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Antoni Font Guiteras, PhD, Study Director — Universitat Autonoma de Barcelona
Locations (1):
- Esther Margarit, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No